CLINICAL TRIAL: NCT02371590
Title: A Phase 2 Clinical Trial To Evaluate Lenalidomide And Obinutuzumab For The Treatment Of Patients With Not Previously Treated Chronic Lymphocytic Leukemia
Brief Title: Lenalidomide and Obinutuzumab for Previously Untreated CLL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study Not Activated Due to Contract Issues
Sponsor: University of California, San Diego (Other)
Collaborators: Celgene Corporation (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Choi, Assistant Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150342/161104
Record Dates: First submitted 2015-02-13; First posted 2015-02-25 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: cancer; lenalidomide; obinutuzumab; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms | interventions — Lenalidomide; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenalidomide-Obinutuzumab (Experimental): All patients receive the combination of lenalidomide and obinutuzumab. There is no randomization or comparator arm.
  Interventions: Drug: Lenalidomide; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide is administered orally once daily on Days 8-28 of each 28 day cycle. The starting dose for all patients is 5 mg PO daily. At the start of each cycle, there is intra-patient dose-escalation to a maximum of 25mg daily, as tolerated.
  The study consists of a 6 month treatment period with obinutuzumab and lenalidomide, and an indefinite period of treatment with lenalidomide for as long as it is helpful and tolerated by subject.
  Other Names: Revlimid
Drug: Obinutuzumab — Obinutuzumab is administered as follows: Cycle 1: 100mg IV on day 1, 900 mg IV on day 2, 1000mg day 8, 1000 mg on day 15. Cycles 2-6: 1000mg IV on day 1.
  Other Names: Gazyva

SUMMARY:
This is phase 1/2 study for patients with CLL or (SLL) who have not been previously treated. This study will evaluate whether obinutuzumab and lenalidomide is safe and tolerable in this setting and induce complete clinical responses.

DETAILED DESCRIPTION:
This is phase 1/2 study for patients with CLL or (SLL) who have not been previously treated. The primary endpoint is to determine safety and tolerability of the regimen and determine complete response (CR) to therapy. The secondary endpoints will assess the impact of treatment on progression free and overall survival

Eligible patients will receive obinutuzumab for 6 x 28 day cycles. Patients will also receive lenalidomide orally once daily on days 8-28 of each 28 day cycles. The starting dose for all patients is 5 mg PO daily. At the start of each cycle, there is intra-patient dose-escalation to a maximum of 25mg daily, as tolerated.

ELIGIBILITY:
* Main Inclusion Criteria:

  1. Clinical and phenotypic verification of B cell CLL or SLL and measurable disease.
  2. Prior therapy: no prior CLL therapy.
  3. Patients must have progressive disease based on 2008 iwCLL definition with one of the following:
* Symptomatic or progressive splenomegaly
* Symptomatic lymph nodes, nodal clusters, or progressive lymphadenopathy
* Progressive anemia (hemoglobin ≤ 11 g/dL)
* Progressive thrombocytopenia (platelets ≤ 100 x 109/L)
* Weight loss > 10% body weight over the preceding 6 month period
* Fatigue attributable to CLL
* Fever or night sweats for > 2 weeks without evidence of infection
* Progressive lymphocytosis with an increase of > 50% over a 2-month period or an anticipated doubling time of less than 6 months.
* Able to take aspirin (81mg or 325mg) daily, warfarin, low molecular weight heparin, or equivalent anticoagulation as prophylactic medication.
* All study participants must be registered into the mandatory Revlimid REMS program, and be willing and able to comply with the requirements of REMS.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours prior to starting Revlimid and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control.
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS program.
* ECOG performance status of 0-2.
* Adequate hematologic function
* Adequate renal function
* Adequate hepatic function

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies. Women for child-bearing age must obtain a pregnancy test and pregnant or breast feeding females are excluded.
* Known hypersensitivity to thalidomide or lenalidomide (if applicable), including development of erythema nodosum or a desquamating rash while taking thalidomide or similar drugs.
* Deep vein thrombosis or superficial thrombophlebitis of any cause on current anticoagulation therapy at the time of screening.
* Patients who are currently receiving another investigational agent are excluded.
* Current infection requiring parenteral antibiotics.
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV); or known active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV) based on detectable viral load. Patients who are seropositive because of hepatitis B virus vaccine or passive immunization by intravenous immunoglobulin (IVIG) are eligible.
* Active malignancy within the previous 2 years (other than completely resected non-melanoma skin cancer or carcinoma in situ).
* Known central nervous system (CNS) involvement by malignancy.
* Untreated autoimmunity such as autoimmune hemolytic anemia, or immune thrombocytopenia.
* Insufficient recovery from surgical-related trauma or wound healing.
* Impaired cardiac function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose limiting toxicity | 1 year
  For phase 1 portion of study
Complete Response Rate | 2 years
  For phase 2 portion of study: iwCLL 2008 defined complete response rate

SECONDARY OUTCOMES:
Number of patients with adverse events associated with lenalidomide-obinutuzumab | 2 years
Progression free survival rate | 2 years
  Progression free survival rate at completion of combination therapy, total progression free survival, and overall survival determined by International Working Group in CLL (iwCLL) criteria
Overall response rate | 2 years
  Overall response rate (Complete response + partial response) and stable disease rate (also based on 2008 iwCLL guidelines), also at the time of primary endpoint response assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Choi, MD, Principal Investigator — UC San Diego Moores Cancer Center
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States